## CONSENT FORM FOR PATIENTS/ VOLUNTEERS IN CLINICAL RESEARCH PROJECT

EXercise TheRApy in Mesothelioma - A Feasibility Study

## EXTRA-Meso Feasibility Study

## **Informed Consent Form**

Chief investigator: Dr Selina Tsim Patient Study ID Number: \_\_\_\_\_ Please Initial 1. I confirm that I have read and understand the information sheet dated ...... (Version .....) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. 2. I agree that I have had the opportunity to ask questions about the study and that these questions have been answered satisfactorily. 3. I agree that my participation is completely voluntary and that I am free to withdraw at any time, without giving a reason, without my medical care or legal rights being affected. 4. I agree to data collected about me being published as part of a research project. My identity will not be revealed in any publication. 5. I agree to relevant sections of my clinical records being accessed by the research team in order to collect data as part of the study. 6. I understand the study involves random allocation of treatment, which neither myself nor the researchers can influence. 7. I agree to the recording of my measurements of fitness, as described in the Patient Information Sheet. 8. I agree to the recording of my quality of life and symptom questionnaire results, as described in the Patient Information Sheet. 9. I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from NHS Greater Glasgow and Clyde (study sponsor), where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. 10. I consent to my GP being informed of my participation in this study.

| 11. I give permission for n<br>Index (CHI) number to be | | and NHS or Community Health<br>ourposes |
|---|---|---|
| 12. I understand that the other research in the future researchers. | | out me will be used to support nonymously with other |
| 13. I agree to take part in | the study. | |
| Optional | | |
| up to an hour and will be | audio recorded. I under | erstand that the interview will last stand that the interviews will be once this has taken place. |
| 15. I agree to anonymised qu | uotes being used in poss | sible publications. |
| Please sign and date l | below. | |
| ame of Participant | Date | Signature |
| ame of researcher | Date | Signature |
| For completion by person to | aking consent: | |
| Please <b>initial</b> the box if cor | nsent was undertaken re | emotely |
| <u>-</u> | | ticipant, 1 original for the e patient's clinical notes. |
| | | copy of the study results and we will mail this to you: |
| Postal address or ema | il address: | |
| | | _ |